CLINICAL TRIAL: NCT06802159
Title: A Comparative Analysis of Methods for Rehabilitation of Unilateral Spatial Neglect (USN) in Stroke Patients: Conventional Therapy, Computerized Cognitive Training and Eye Movement Biofeedback Training
Brief Title: Rehabilitation Methods for Unilateral Spatial Neglect in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health (Other)
Responsible Party: Principal Investigator, Mikhail Soldatov, Dr, Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NeglectRehab01
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Unilateral Spatial Neglect (USN)
Keywords: Unilateral spatial neglect; stroke; rehabilitation; eye-tracking; computerized cognitive training
MeSH Terms: conditions — Stroke | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional group (Active Comparator): Patients with prescribed traditional neuropsychological rehabilitation. The rehabilitation program consisted of 6-10 sessions. On average, one session lasted 25-30 minutes, which was also limited by inpatient conditions (no correctional sessions with a neuropsychologist longer than 30 minutes) and the patient's fatigue.
  Interventions: Behavioral: Conventional therapy
- Eye tracker group (Experimental): Patients with assigned rehabilition to the alternative communication device - oculograph C Eye Pro (Assistech). The correctional program consisted of 6-10 sessions. On average, one session lasted 25-30 minutes, which was also limited by inpatient conditions (no correctional sessions with a neuropsychologist longer than 30 minutes) and patient fatigue.
  Interventions: Behavioral: Eye tracking based therapy
- Cognitive training group (Experimental): Patients with assigned rehabilitation on the RehaCom modular therapy system (HASOMED GmbH;). The rehabilitation program consisted of 6-10 sessions. One session lasted 25-30 minutes, which was also limited by inpatient conditions (no correctional sessions with a neuropsychologist longer than 30 minutes) and the patient's fatigue.
  Interventions: Behavioral: Cognitive therapy

INTERVENTIONS:
Behavioral: Conventional therapy — The methods of traditional neuropsychological rehabilitation used in the classes included:
  * attention tasks: proofreading tests, Schulte's Table;
  * spatial thinking tasks: copying, drawing, tasks using Nikitin cubes;
  * text reading tasks: texts from the Luria album. Each session began with oculomotor exercises. The correction programs differed by the type of feedback given to the patient in the course of correction.
  Feedback in this type of intervention is in the form of prompts from a specialist.
  Arms: Conventional group
Behavioral: Eye tracking based therapy — Rehabilitation in this group was carried out using an alternative communication device - oculograph C-Eye Pro (Assistech). The use of the device is characterized by a number of features: the presence of the eye movement biofeedback function (the patient and the specialist can see where the patient's gaze is directed by the movement of the red dot on the screen), the device needs to be pre-calibrated before the beginning of the session. To implement rehabilitation activities such tasks were used as:
  * Visual field training;
  * Word composing;
  * Vowel insertion;
  * Reading;
  * etc. The peculiarity of correction on the apparatus of alternative communication - oculograph - was the use of visual biological communication, visual biological communication, also in case of wrong answer a sound signal followed.
  Arms: Eye tracker group
Behavioral: Cognitive therapy — Rehabilitation of patients in the second experimental group was carried out on the RehaCom modular therapeutic system. The modular system includes a dedicated keyboard that has: numbers 1-9, 4 ok buttons, 4 arrow buttons, 2 pause/tip buttons and 2 exit/cancel buttons. Most of the tasks are performed using the keyboard, some of the tasks involved touch screen control. Tasks with stimulus images in the left screen space were used for rehabilitation activities:
  * "Saccades";
  * "Attention and Concentration";
  * "Planar Imagination";
  * "General Presentation and Reading";
  * "Shopping";
  * "Daily routine". A feature of the correction on the modular therapy system was the involvement of a motor component, playing a sound cue or visual cue when an error occurred.
  Arms: Cognitive training group

SUMMARY:
Stroke remains one of the leading causes of mortality and disability worldwide. Between 30% and 40% of patients who have had an acute cerebral hemorrhage, develop unilateral spatial neglect syndrome (USN).

USN is observed in 24% of patients with left-hemispheric stroke and 45% of patients with right-hemispheric lesions in the acute phase acute phase and in 20% of patients in the chronic phase.

The presence of USN significantly complicates the rehabilitation process and negatively affects the functional outcomes. The complexity of USN correction is due to the heterogeneity of its manifestations and combination with other cognitive disorders. In 30-50% of patients with USN anosognosia is observed, in 60% - memory and attention disorders.

Traditional methods of rehabilitation lead to significant improvement in 30-50% of patients with USN. The use of combined methods of treatment, including pharmacotherapy and non-medication methods, can improve efficacy by up to 70-80%. This indicates the need to develop and investigate new approaches to correct USN.

Despite the growing number of studies in this area, there is still no unified approach to selecting the optimal method of USN correction for each individual patient.

Different methods of rehabilitation may have different effects on neuroplasticity processes, which opens new perspectives for optimization of rehabilitation strategies.

DETAILED DESCRIPTION:
Stroke remain one of the leading causes of death and disability worldwide. According to the World Health Organization, about 15 million cases of stroke are registered annually, of which 5 million are fatal and another 5 million result in permanent disability.

In Russia, about 450 thousand cases of stroke are registered annually, with a mortality rate of about 35% during the first year after stroke. The frequency of ischemic strokes is 80-85%, hemorrhagic strokes - 15-20%.

According to the localization of the lesion, strokes in the middle cerebral artery basin are the most common (up to 50-60% of cases), followed by strokes in the vertebrobasilar basin (20-25%) and the anterior cerebral artery basin (10-15%).

Disability after a stroke is observed in 70-80% of surviving patients, with about 20-30% requiring constant nursing care.

Neuro-ophthalmologic disorders develop in 40-60% of cases in patients who have undergone stroke, while sensory inattention develops in 30-40% of cases. Sensory inattention, or neglect syndrome, is a manifestation of optic-spatial gnostic disorders.

In a systematic review analyzing the incidence of neglect syndrome after stroke, Esposito et al. reported that the syndrome occurs in 24%-with left hemispheric brain damage and 45% of patients with right hemispheric brain damage in the acute phase and in 20% 5 of patients in the chronic phase, but the prevalence of neglect syndrome varies between studies (up to 82%).

The scientific relevance of the study on the topic " A Comparative Analysis of Methods for Rehabilitation of Unilateral Spatial Neglect (USN) in Stroke Patients: Conventional Therapy, Computerized Cognitive Training and Eye Movement Biofeedback Training" is due to the high prevalence and significant impact of this syndrome on the rehabilitation process and quality of life of patients after stroke.

Unilateral spatial neglect (USN) is one of the most frequent and disabling syndromes in stroke, especially when the right hemisphere is affected. According to various studies, the prevalence of USN among stroke patients ranges from 13% to 81%. This wide range is due to differences in diagnostic methods and timing of evaluation after stroke. In the acute phase (first 2 weeks), USN is observed in 85% of patients with right hemispheric stroke, and 3 months after stroke, symptoms persist in 36% of patients.

The presence of USN significantly complicates the rehabilitation process and negatively affects functional outcomes. Studies show that patients with USN have a longer hospitalization period (28 days longer on average) compared to patients without USN. In addition, patients with USN are 20-40% less likely to achieve independence in activities of daily living. This leads to a significant increase in the economic burden: the presence of USN increases the cost of care for a patient after stroke by 25-40%.

The complexity of USN correction is due to the heterogeneity of its manifestations and its frequent combination with other cognitive disorders. Anosognosia (denial of their disease) is observed in 30-50% of patients with USN, and about 60% of patients have concomitant disorders of memory and attention. These factors make it difficult to involve patients in the rehabilitation process and require an individualized approach to the choice of correction methods.

Traditional rehabilitation methods lead to meaningful improvement in 30-50% of patients with USN. However, the use of combined treatment methods, including pharmacotherapy and non-medication methods, can increase the effectiveness to 70-80%. This indicates the need for the development and research of new approaches to the correction of USN.

In recent years, innovative methods for the correction of USN, such as the use of virtual reality and noninvasive brain stimulation, have been actively developed. The use of virtual reality can significantly improve the rehabilitation outcomes of patients with USN.

Currently, computerized training methods are very popular for improving cognitive functions, which include many tasks in various domains: memory, attention, perception, thinking, executive functions, etc. Similar computer solutions, for example RehaCom, can also be used to rehabilitate USN. In addition to the above functions, tasks in this software include training of visual functions, including scanning of affected visual fields, etc. On the other hand, it is extremely promising to use the method of training eye movements to study the affected hemifield in patients with USN. To provide biological feedback, this training uses the eye tracking method. This is a non-invasive method that allows even patients with paresis to work with rehabilitation equipment.

However, despite the growing number of studies in this area, there is still no unified approach to selecting the optimal method of USN correction for each specific patient. Existing studies often have methodological limitations and insufficient statistical power, which makes it difficult to formulate unambiguous recommendations.

In addition, most studies focus on the short-term effects of rehabilitation, whereas data on long-term outcomes are limited. According to some estimates, in 10-15% of patients with USN, symptoms persist for more than a year after stroke, which emphasizes the need to study the long-term effects of different methods of correction.

The relevance of comparative analysis of methods of USN correction is also due to the growing understanding of brain neuroplasticity and its role in stroke recovery. Studies show that different rehabilitation methods can differentially affect neuroplasticity processes, which opens new perspectives for optimizing rehabilitation strategies.

Finally, it is important to note that USN is often combined with other post-stroke disorders such as aphasia, apraxia and motor disorders. This requires an integrated approach to rehabilitation and the study of the interaction of different methods of correction.

Thus, the scientific relevance of the comparative analysis of methods of correction of USN in patients with stroke is due to the high prevalence of the syndrome, its significant impact on the rehabilitation process and quality of life of patients, as well as the need to develop more effective and personalized approaches to treatment. Such a study can make a significant contribution to the optimization of rehabilitation strategies and improvement of functional outcomes in patients with post-stroke USN.

ELIGIBILITY:
Inclusion Criteria:

* Normal cognitive development in accordance with age and educational level;
* diagnosis with codes I63, I61 (ICD);
* presence of unilateral spatial neglect syndrome in the neuropsychological status.

Exclusion Criteria:

* presence of mental and somatic pathology of severe degree and in decompensation stage;
* the presence of gross oculomotor disorders;
* presence of a sensory visual defect of moderate to severe severity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual search for objects in the left and right hemifield among distractors | Measurement compared to baseline after 2 weeks
  The visual search task is aimed at determining the latent search time for subject images (soccer ball, blue suitcase, potatoes in a glass) among a large number of distractors. The test is also performed on a C-Eye II Pro. The test procedure starts with recalibration, with a total of 5 calibration points. The test utilizes the visual biofeedback function - the specialist and the subject can observe the gaze movement of the patient. At the Measurement compared to baseline after 2 weeks beginning of the test, the patient is asked to scrutinize the appeared picture (target and distractor images appear on the screen at the same time) for 30 seconds. After that, the patient should fix his or her gaze on the image of a white question mark in the center of the screen. Next, search tasks are given to find: soccer ball, red felt-tip pen, blue suitcase, green light bulb, planet earth, fries in a glass. The patient's task was to find all target objects in less than 25 seconds from a fixed point.

SECONDARY OUTCOMES:
Albert test | Measurement compared to baseline after 2 weeks
  The line-drawing test aims to estimate the latent search time of stimuli, to quantify the missed stimuli according to their location on the sheet. The test involves the presentation of a sheet with 40 lines, 2.5 minutes long, organized in 6 rows of 6 lines and one row of 5 lines. Accordingly, there are 18 lines on the right and left and 5 on the left. The patient's task is to cross out all the lines as quickly as possible (after 5 minutes the test is interrupted). Processing of the test results: the maximum number of points is 41, which means that the examinee found all the bells. Indicative in interpreting the results of parameter tests is the percentage of line skips in the left half of the sheet from the total number of skips. Thus, if more than 70% are recorded, we can assume the development of visual inattention
Bell's Test | Measurement compared to baseline after 2 weeks
  The is aimed at estimating the latent search time of stimuli, at quantifying the missed stimuli depending on their location on the sheet. An important feature of the test is the presence of distractors in the stimulus material. Initially, the subject is presented with a "demonstration" sheet containing an enlarged version of each of the distractors and one circled bell. As part of the test, a sheet showing a large number of small black images is presented, among which 35 bells are distributed in 7 columns. In total there are 3 columns on the right and left and one in the center. The patient's task is to cross out all the bells as quickly as possible. Processing of the test results: the maximum number of points is 35, which means that the subject found all the bells. If the patient makes more than 3 omissions, we can talk about possible attention deficit, but if the number of omissions is more than 6, it indicates signs of visual inattention.
Line bisection test | Measurement compared to baseline after 2 weeks
  The test is aimed at determining the degree of displacement of the subjective center. The test involves the presentation of 20 horizontal lines of different lengths. The first and last lines are demonstration lines, on which the specialist demonstrates the instruction and independently places a vertical mark in the center of each line. The 18 stimulus lines are divided into three blocks according to their location on the sheet: 6 on the left, in the center and on the right. The task of the test subject is to mark the center on each of the lines. The test results were processed according to the formula proposed by Schenkenberg to get the % offset of the center mark. A negative value indicates a leftward shift, a positive value indicates a rightward shift Interpretation. The left and center lines are significant for the analysis. Thus, if the mean value for left line blocks is > 7% and for center line blocks > 5%, we can assume the development of neglect syndrome
Test of complex competitive stimulation in both visual hemifields | Measurement compared to baseline after 2 weeks
  The test is aimed at determining the latent search time of stimuli located in both visual fields among distractors. The test is performed on C-Eye II Pro. The test utilizes the visual biofeedback function - the technician and the subject can observe the gaze movement of the patient. As part of the test, the test taker is initially presented with a demonstration sheet depicting all of the figures demonstrated in the test. The subject is asked to name only one figure, for a total of 8 figures. Then there are 12 presentations of figures in different numbers and positions relative to each other: no less than 1 and no more than 3 figures are displayed on the screen at the same time, before each presentation the patient is shown a blue circle located in the center. The patient's task is to find the figures on the screen, look at them, and name them. If the subject searches for a figure for longer than 25 seconds, the specialist proceeds to the next presentation.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Federal Center of Brain and Neurotechnologies of the FMBA of Russia, Moscow, Moscow
  - Federal Center of Brain and Neurotechnologies of the FMBA of Russia, Moscow

IPD SHARING:
Plan to Share IPD: No
Only on special request